CLINICAL TRIAL: NCT03896789
Title: Implementation Fidelity and Benefits of the Critical Care Pediatric Guideline Adherence and Outcomes Program in Traumatic Brain Injury
Brief Title: Pediatric Guideline Adherence and Outcomes- Argentina
Acronym: PEGASUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Children's National Research Institute (Other); Centro de Informática e Investigación Clínica (CIIC) (Unknown); Washington State University (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Monica Vavilala, Professor, School of Medicine: Anesthesiology and Pain Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00005629; 1R01NS106560-01A1 (NIH)
Record Dates: First submitted 2019-01-07; First posted 2019-04-01 (Actual); Results first posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: TBI (Traumatic Brain Injury)
Keywords: guideline adherence; implementation fidelity; pediatric
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: Parallel cluster randomized cluster trial (RCT) following a baseline data collection period when all sites are in the 'control/usual care state'.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care, then Usual Care (Control) (No Intervention): All sites will collect usual care data during the baseline and post-randomization study periods. This arm (half of the sites) will maintain usual care. They will receive the opportunity for the PEGASUS program training (intervention) at the end of study.
- Usual Care, then PEGASUS Program (Intervention) (Experimental): All sites will collect usual care data during the baseline study period. With intention-to-treat, after randomization, this arm (half of the sites) will be considered experimental and receive intervention training and then deliver the PEGASUS program (intervention) along with other Usual Care.
  Interventions: Other: PEGASUS Program for Care

INTERVENTIONS:
Other: PEGASUS Program for Care — This is in essence a checklist of pediatric guidelines to follow for participants who meet inclusion criteria. Site staff will receive training in how to implement this pathway into their usual care.
  Arms: Usual Care, then PEGASUS Program (Intervention)

SUMMARY:
Pediatric traumatic brain injury (TBI) is the leading killer of children worldwide but effective treatments for TBI are limited. Although evidenced-based pediatric TBI guidelines exist, adherence to these guidelines is low,leading us to develop a new Pediatric Guideline Adherence and Outcomes (PEGASUS) program to increase TBI guideline adherence. We propose to test the PEGASUS program's ability to improve TBI guideline adherence and outcomes.

DETAILED DESCRIPTION:
Specific Aim 1: Determine the relationship between PEGASUS program implementation and TBI guideline adherence (Aim 1a), and assess system, provider, patient, implementation and guideline factors associated with TBI guideline adherence (Aim 1b). Hypothesis: Centers that receive the PEGASUS program have higher TBI guideline adherence (main outcome), as well as better discharge survival and 3-month Glasgow Outcome Scale-Extended (GOSE) score (secondary outcomes) than centers who receive usual care.

Specific Aim 2: Create a value stream map (VSM) to identify value-added processes of care associated with TBI guideline adherence. Hypothesis: ICU activity flows of TBI care during the first 72 hours will reveal value-added as well as non-value-added processes in severe TBI care. PEGASUS program implementation will result in more value-added TBI care processes and better TBI guideline adherence.

Specific Aim 3: Use computer simulation to develop and disseminate a real-world best practices blueprint for TBI guideline adherence. Hypothesis: This model will identify the impact of the PEGASUS program on key performance indicators (KPIs), outcomes (Aim 1), and process activities (Aim 2). Iterative computer simulations will then demonstrate the relationship among PEGASUS program components and how relative changes in these components impact the magnitude, direction and choice of operations downstream in TBI care and patient outcomes to inform development of a blueprint for wide dissemination of best-practice guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Mechanism or head CT consistent with TBI
* <18 years old
* Glasgow Coma Scale (GCS) score ≤8 at any point during hospital admission, motor GCS≤5 if intubated

Exclusion Criteria:

- none

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 505 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2023-09-26 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Monica Vavilala, MD, Principal Investigator — University of Washington
Locations (16):
- Argentina (14):
  - Hospital Sor Ludovica, La Plata, Buenos Aires
  - Hospital Interzonal Especializado Materno Infantil, Mar del Plata, Buenos Aires
  - Hospital el Cruce, San Juan Bautista, Buenos Aires
  - Hospital Municipal del Nino de San Justo, San Justo, Buenos Aires
  - Hospital de Ninos Eva Peron, Catamarca, Catamarca Province
  - Hospital Materno Infantil Dr. Hector Quintana, San Salvador de Jujuy, Jujuy Province
  - Hospital Regional Reconquista, Reconquista, Santa Fe Province
  - Hopital Victor J. Vilela, Rosario, Santa Fe Province
  - Hospital del Nino Jesus, San Miguel de Tucumán, Tucumán Province
  - Hospital de La Santisima Trinidad, Córdoba
  - Hospital Humberto Notti, Mendoza
  - Hospital Publico Materno Infantil, Salta
  - Hospital Alassia, Santa Fe
  - Centro Provincial de Salud Infantil Eva Peron, Santiago del Estero
- Hospital Carlos Van Buren, Valparaíso, Chile
- Hospital de Trauma Manuel Giagni, Asunción, Paraguay

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared with Co-Investigators
Supporting Information: ICF
Time Frame: Monthly as available

REFERENCES:
- [Derived] Velonjara J, Mills B, Lujan S, Petroni G, Bell MJ, Guadagnoli N, Mock C, Hughes JP, Vavilala MS, Rowhani-Rahbar A; PEGASUS Argentina Study Group. The Pediatric Guideline Adherence and Outcomes (PEGASUS Argentina) program in severe traumatic brain injury: study protocol adaptations during the COVID-19 pandemic for a multisite implementation-effectiveness cluster randomized controlled trial. Trials. 2022 Dec 5;23(1):980. doi: 10.1186/s13063-022-06938-x. PMID 36471399

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were screened based on ICU admission at 16 South American study hospitals between September 1, 2019 and September 30, 2023. The first participant was enrolled on September 9, 2019 and the last participant was enrolled September 26, 2023.
Pre-assignment Details: Due to COVID-19, we reverted to a parallel-cluster design before randomization, resulting in a baseline period (9/1/19-7/13/20) with usual care data collected at all sites. Arm assignment and site notification was 7/13/20. Participants enrolled between 7/14/20-9/30/20 during intervention site training are included in the assigned arm (intention-to-treat) due to possible behavior change once assignment was known. Intervention implementation began for participants enrolled between 10/1/20-9/30/23.
Units Other Than Participants: Sites
Groups:
- Usual Care, Then Usual Care (Control): All sites collected usual care data from participants enrolled before randomization. This arm (8 sites) was randomized to maintain usual care (control) on 7/13/2020. Participants recruited post-randomization are included in the post-randomization period. They will receive the opportunity for the PEGASUS program training (intervention) after the end of study.
- Usual Care, Then PEGASUS Program (Intervention): All sites collected usual care data from participants enrolled before randomization. This arm (8 sites) was randomized to receive the PEGASUS program (intervention) on 7/13/2020. Intervention site training occurred before the intervention was implemented for new participants beginning 10/1/2020. Participants recruited post-randomization but pre-implementation are included in the post-randomization period through end of recruitment 9/30/2023.
  PEGASUS Program for Care: This is in essence a checklist of pediatric guidelines to follow for participants who meet inclusion criteria. Site staff will receive training in how to implement this pathway into their usual care.
Period: Baseline
Arm/Group | Usual Care, Then Usual Care (Control) | Usual Care, Then PEGASUS Program (Intervention)
Started | 55; 8 Sites | 61; 8 Sites
3-month Post-admission Follow-up | 52; 8 Sites (3 participants died in-hospital, so had no 3-month follow-up.) | 55; 8 Sites (6 participants died in-hospital, so had no 3-month follow-up.)
Completed | 51; 8 Sites | 53; 8 Sites
Not Completed | 4; 0 Sites | 8; 0 Sites
Not completed — Lost to Follow-up | 1 | 2
Not completed — Death | 3 | 6
Period: Post-Randomization
Arm/Group | Usual Care, Then Usual Care (Control) | Usual Care, Then PEGASUS Program (Intervention)
Started | 208; 8 Sites (No participants contribute to both Baseline and Post-Randomization periods. All participants in the Post-Randomization period are new participants who were admitted and enrolled after the site randomization. All participants in this arm received usual care.) | 181; 8 Sites (No participants contribute to both Baseline and Post-Randomization periods. All participants in the Post-Randomization period are new participants who were admitted and enrolled after site randomization. Participants in this arm received usual care during the Baseline Period. Post-Randomization participants were assigned intention-to-treat; participants enrolled during site training were included along with those after implementation who received usual care and the PEGASUS intervention.)
3-month Post-admission Follow-up | 196; 8 Sites (12 participants died in-hospital, so had no 3-month follow-up.) | 168; 8 Sites (13 participants died in-hospital, so had no 3-month follow-up.)
Completed | 184; 8 Sites | 157; 8 Sites
Not Completed | 24; 0 Sites | 24; 0 Sites
Not completed — Lost to Follow-up | 12 | 11
Not completed — Death | 12 | 13

BASELINE CHARACTERISTICS:
Population: 16 sites contributed participants during baseline period. After randomization, 8 of those sites were assigned Control and 8 were assigned Intervention. Participants were allocated to the study arms based on their admission to either the control study hospitals or intervention study hospitals.
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care, Then Usual Care (Control) | Usual Care, Then PEGASUS Program (Intervention) | Total
Number analyzed (Participants) | 263 | 242 | 505
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The two row titles encompass two participant recruitment periods with patients participating in only one period. The sum of the rows equals the overall.
  Participants enrolled during baseline (study start through randomization on 7/13/20) provided usual care data.
  Participants enrolled during post-randomization (beginning 7/14/20 through study end) provided either usual care or intervention implementation data. This period was the population used in the primary analysis.
  years
    Baseline: number analyzed (Participants) | 55 | 61 | 116
    Baseline | 6.2 (4.7) | 7.7 (5.7) | 7.0 (5.3)
    Post-Randomization: number analyzed (Participants) | 208 | 181 | 389
    Post-Randomization | 6.9 (4.5) | 7.8 (4.8) | 7.3 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The two row titles encompass two participant recruitment periods with patients participating in only one period. The sum of the rows equals the overall.
  Participants enrolled during baseline (study start through randomization on 7/13/20) provided usual care data.
  Participants enrolled during post-randomization (beginning 7/14/20 through study end) provided either usual care or intervention implementation data. This period was the population used in the primary analysis.
  Participants
    Baseline: number analyzed (Participants) | 55 | 61 | 116
    Baseline: Female | 19 | 23 | 42
    Baseline: Male | 36 | 38 | 74
    Post-Randomization: number analyzed (Participants) | 208 | 181 | 389
    Post-Randomization: Female | 77 | 58 | 135
    Post-Randomization: Male | 131 | 123 | 254
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Total Glasgow Coma Scale (GCS) score <=8 [Count of Participants; unit: Participants] — GCS score extracted from patient medical record as assessed by a provider. Used to measure changes in consciousness, including coma. The total score is made up of the sum of three components: eye response (1-4), verbal response (1-5), and motor response (1-6). The range is 3-15, with 15 being fully responsive in all component categories and 3 being fully non-responsive in all categories. A score less than or equal to 8 is typically classified as a severe traumatic brain injury when used in connection with a head injury. Population: The two row titles encompass two participant recruitment periods with patients participating in only one period. The sum of the rows equals the overall.
  Participants enrolled during baseline (study start through randomization on 7/13/20) provided usual care data.
  Participants enrolled during post-randomization (beginning 7/14/20 through study end) provided either usual care or intervention implementation data. This period was the population used in the primary analysis.
  Participants
    Baseline: number analyzed (Participants) | 55 | 61 | 116
    Baseline: At admission <=8 | 35 | 48 | 83
    Baseline: Deteriorated <=8 | 18 | 13 | 31
    Baseline: Total GCS >8 (but motor<=5) | 2 | 0 | 2
    Post-Randomization: number analyzed (Participants) | 208 | 181 | 389
    Post-Randomization: At admission <=8 | 146 | 138 | 284
    Post-Randomization: Deteriorated <=8 | 62 | 43 | 105
    Post-Randomization: Total GCS >8 (but motor<=5) | 0 | 0 | 0
Any extracranial injury [Count of Participants; unit: Participants] — Non-head Abbreviated Injury Scale (AIS) score >0 indicates extracranial injury (1-6). Non-head AIS score=0 indicates isolated TBI (0).
  AIS is a scale assessing injury severity for different body regions, 0=uninjured, 1=minor to 6=unsurvivable. Non-head AIS is the highest value of any non-head region AIS. Population: The two row titles encompass two participant recruitment periods with patients participating in only one period. The sum of the rows equals the overall.
  Participants enrolled during baseline (study start through randomization on 7/13/20) provided usual care data.
  Participants enrolled during post-randomization (beginning 7/14/20 through study end) provided either usual care or intervention implementation data. This period was the population used in the primary analysis.
  Participants
    Baseline: number analyzed (Participants) | 55 | 61 | 116
    Baseline: No | 20 | 19 | 39
    Baseline: Yes | 35 | 42 | 77
    Post-Randomization: number analyzed (Participants) | 208 | 181 | 389
    Post-Randomization: No | 61 | 31 | 92
    Post-Randomization: Yes | 147 | 150 | 297
Injury Severity Scale (ISS) [Mean (Standard Deviation); unit: units on a scale] — ISS range (0-75) The sum of the square of the highest three body region Abbreviated Injury Scale (AIS) scores. AIS range is 0-6, with 0=uninjured, 1=minor to 6=unsurvivable. If any body region has AIS=6, then ISS=75, regardless of other body region AIS scores. Higher score indicates higher total injury severity. Population: The two row titles encompass two participant recruitment periods with patients participating in only one period. The sum of the rows equals the overall.
  Participants enrolled during baseline (study start through randomization on 7/13/20) provided usual care data.
  Participants enrolled during post-randomization (beginning 7/14/20 through study end) provided either usual care or intervention implementation data. This period was the population used in the primary analysis.
  units on a scale
    Baseline: number analyzed (Participants) | 55 | 61 | 116
    Baseline | 26.9 (20.8) | 28.8 (18.7) | 27.3 (20)
    Post-Randomization: number analyzed (Participants) | 208 | 181 | 389
    Post-Randomization | 26.3 (18.8) | 29.6 (16.7) | 27.8 (17.9)

OUTCOME MEASURES:

1. Primary Outcome: First 3-day Cumulative Intensive Care Unit (ICU) Traumatic Brain Injury (TBI) Guideline Adherence Rate, Overall
Description: Adherence to nine of the 15 Brain Trauma Foundation TBI guideline indicators were determined for indicators that were logistically relevant in the South American clinical care context.
  To determine the first 3-day cumulative ICU TBI guideline adherence rate, adherence to each indicator was first determined for each participant and coded as yes/no/not applicable for each day. For continuous indicators, the daily guideline adherence rate to each indicator was averaged over the first three days. For non-continuous indicators, the daily guideline adherence rate to each indicator was defined as 100% if adherence was achieved within any of the first three days. The 3-day cumulative ICU TBI guideline adherence rate, overall was determined by averaging adherence rates across all nine guideline indicators. Guideline adherence was clustered by site and grouped by site allocation (control or intervention).
Time Frame: ICU Stay for severe TBI care, first 3 days from admission (or until death or discharge, if before 3 days).
Population: We compared control and intervention arms post-randomization (07/13/20) in statistical analysis. Baseline period data contributed to other adjusted analyses.
Measure: Mean (Standard Deviation); unit: mean percentage of guideline adherence
Arm/Group | Usual Care, Then Usual Care (Control) | Usual Care, Then PEGASUS Program (Intervention)
Number analyzed (Participants) | 263 | 242
mean percentage of guideline adherence
  Baseline: number analyzed (Participants) | 55 | 61
  Baseline | 81.7 (12.9) | 81.0 (13.2)
  Post-Randomization: number analyzed (Participants) | 208 | 181
  Post-Randomization | 83.7 (11.5) | 84.4 (12.8)
Statistical Analysis 1: Comparison: Usual Care, Then Usual Care (Control) vs Usual Care, Then PEGASUS Program (Intervention); Null hypothesis: Assuming no difference between usual care (control) and PEGASUS (intervention). We used 2011-2012 results from prior pilot work in Argentina (58.6% TBI guideline adherence) to determine a sample size of 432 eligible patients (216 per arm) for the planned parallel cluster RCT, which would have 80% power to detect a 18.7% higher ICU TBI guideline adherence rate with programme implementation, with a two-sided alpha of 5%, and an intraclass coefficient of 0.05; Test type: Superiority; p = .95, Mixed Models Analysis — The primary outcome was analyzed using a multi-level mixed-effects model, which included a random effect for site (to account for potential provider clustering) and fixed effects for covariates; Included covariates were age, gender, head maximum AIS, non-head maximum AIS, nurse: patient ratio and baseline TBI guideline adherence scores; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-3.3 to 3.5]

2. Secondary Outcome: Clinical Pathway Adoption
Description: This outcome will be measured as yes/no for each participant at intervention sites to assess intervention delivery. In essence, the intervention started (use of PEGASUS program clinical pathway) within 24 hours of their eligibility and enrollment.
  Due to our intention-to-treat analysis plan, participants who enrolled after randomization but before intervention implementation at intervention sites are included in the analysis. Although they could not have implemented the intervention, sites were aware of their allocation status and were preparing and training during this interval.
Time Frame: Started within 24 hours of patient eligibility (at admission or deterioration)
Population: Analysis was intention-to-treat. Patients enrolled to the intervention arm after randomization, but before intervention implementation were still included because site investigators and sites were aware of their arm assignment from that date and could have altered behavior during the training interval before implementation start.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care, Then PEGASUS Program (Intervention)
Number analyzed (Participants) | 181
Participants
  Post-Randomization, Pre-Implementation | 11
  Post-Randomization, Post-Implementation Implemented Clinical Pathway | 170
  Post-Randomization, Post-Implementation Did Not Implement Clinical Pathway | 0

3. Secondary Outcome: Glasgow Outcome Scale (GOS) Score at Discharge
Description: Participants' GOS score at hospital discharge from medical record:
  Death-1 (worse) Vegetative State-2 Severe Disability-3 Moderate Disability-4 Good Recovery-5 (better)
  The timing varies for each participant since the duration of hospitalization depended on the clinical care factors of each individual and could not be controlled by the study.
Time Frame: Assessed at Discharge. This varies for each participant since the duration of hospitalization depended on the clinical care factors of each individual and could not be controlled by the study.
Population: The two row titles encompass two participant recruitment periods with patients participating in only one period. The sum of the rows equals the overall.
  Participants enrolled during baseline (study start through randomization on 7/13/20) provided usual care data.
  Participants enrolled during post-randomization (beginning 7/14/20 through study end) provided either usual care or intervention implementation data. This period was the population used in the primary analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Usual Care (Control): All sites collected usual care data from participants enrolled before randomization. This arm (8 sites) was randomized to maintain usual care (control) on 7/13/2020. Participants recruited post-randomization are included in the post-randomization period. They will receive the opportunity for the PEGASUS program training (intervention) after the end of study.
- PEGASUS Program (Intervention): All sites collected usual care data from participants enrolled before randomization. This arm (8 sites) was randomized to receive the PEGASUS program (intervention) on 7/13/2020. Intervention site training occurred before the intervention was implemented for new participants beginning 10/1/2020. Participants recruited post-randomization but pre-implementation are included in the post-randomization period through end of recruitment 9/30/2023.
  PEGASUS Program for Care: This is in essence a checklist of pediatric guidelines to follow for participants who meet inclusion criteria. Site staff will receive training in how to implement this pathway into their usual care.
Arm/Group | Usual Care (Control) | PEGASUS Program (Intervention)
Number analyzed (Participants) | 263 | 242
Participants
  Baseline: number analyzed (Participants) | 55 | 61
  Baseline: Death (all-cause) | 3 | 6
  Baseline: Vegetative state | 0 | 2
  Baseline: Severe disability | 5 | 4
  Baseline: Moderate disability | 3 | 19
  Baseline: Good recovery | 44 | 30
  Post-Randomization: number analyzed (Participants) | 208 | 181
  Post-Randomization: Death (all-cause) | 12 | 13
  Post-Randomization: Vegetative state | 15 | 9
  Post-Randomization: Severe disability | 18 | 17
  Post-Randomization: Moderate disability | 24 | 42
  Post-Randomization: Good recovery | 139 | 100

4. Secondary Outcome: Discharge Survival
Description: Number of survivors at intervention and control sites (descriptive and not powered for this outcome).
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care, Then Usual Care (Control) | Usual Care, Then PEGASUS Program (Intervention)
Number analyzed (Participants) | 263 | 242
Participants
  Baseline: number analyzed (Participants) | 55 | 61
  Baseline: Died in-hospital | 3 | 6
  Baseline: Survived | 52 | 55
  Post-Randomization: number analyzed (Participants) | 208 | 181
  Post-Randomization: Died in-hospital | 12 | 13
  Post-Randomization: Survived | 196 | 168

5. Secondary Outcome: Glasgow Outcome Scale-Extended, Pediatric Version (GOSE-Peds)
Description: We will examine participants' recovery using GOSE-Peds scores. These were assessed by site study staff either in-person, by telephone, or from medical record approximately 3 months after the admission date.
  Death-8 (worse) Vegetative State-7 Severe Disability lower-6 Severe Disability upper-5 Moderate Disability lower-4 Moderate Disability upper-3 Good Recovery lower-2 Good Recovery upper-1 (better)
Time Frame: 3 months post-admission
Population: 3-month outcome assessment among those who survived (enrolled participants less those who died in-hospital) and reached for follow-up. Lost-to-follow-up noted in Participant Flow.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care (Control) | PEGASUS Program (Intervention)
Number analyzed (Participants) | 235 | 210
Participants
  Baseline: number analyzed (Participants) | 51 | 53
  Baseline: Death | 0 | 0
  Baseline: Vegetative state | 0 | 2
  Baseline: Severe disability-lower | 5 | 8
  Baseline: Severe disability-upper | 7 | 10
  Baseline: Moderate disability-lower | 0 | 1
  Baseline: Moderate disability-upper | 4 | 1
  Baseline: Good recovery-lower | 3 | 4
  Baseline: Good recovery-upper | 32 | 27
  Post-Randomization: number analyzed (Participants) | 184 | 157
  Post-Randomization: Death | 0 | 0
  Post-Randomization: Vegetative state | 6 | 9
  Post-Randomization: Severe disability-lower | 27 | 25
  Post-Randomization: Severe disability-upper | 11 | 17
  Post-Randomization: Moderate disability-lower | 4 | 4
  Post-Randomization: Moderate disability-upper | 9 | 8
  Post-Randomization: Good recovery-lower | 26 | 26
  Post-Randomization: Good recovery-upper | 101 | 68

6. Secondary Outcome: Mortality, 3-Month
Description: We will examine participants' mortality at 3 months post discharge
Time Frame: 3 months post admission
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care (Control) | PEGASUS Program (Intervention)
Number analyzed (Participants) | 235 | 210
Participants
  Baseline: number analyzed (Participants) | 51 | 53
  Baseline: Died | 0 | 0
  Baseline: Survived | 51 | 53
  Post-Randomized: number analyzed (Participants) | 184 | 157
  Post-Randomized: Died | 0 | 0
  Post-Randomized: Survived | 184 | 157

7. Other Pre Specified Outcome: Cumulative First 3-day ICU TBI Guideline Adherence Rate, by Extracranial Injury Status
Description: Adherence to nine of the 15 Brain Trauma Foundation TBI guideline indicators were determined for indicators that were logistically relevant in the South American clinical care context.
  To determine the first 3-day cumulative ICU TBI guideline adherence rate, adherence to each indicator was first determined for each participant and coded as yes/no/not applicable for each day. For continuous indicators, the daily guideline adherence rate to each indicator was averaged over the first three days. For non-continuous indicators, the daily guideline adherence rate to each indicator was defined as 100% if adherence was achieved within any of the first three days. The 3-day cumulative ICU TBI guideline adherence rate, overall was determined by averaging adherence rates across all nine guideline indicators. Guideline adherence was clustered by site and grouped by site allocation (control or intervention).
  Here, we stratified by extracranial injury status (isolated TBI vs. TBI and ext
Time Frame: ICU Stay for severe TBI care, first 3 days from admission (or until death or discharge, if before 3 days).
Population: We compared control and intervention arms post-randomization (07/13/20) in statistical analysis by extracranial injury status.
Measure: Mean (Standard Deviation); unit: mean percentage of guideline adherence
Arm/Group | Usual Care, Then Usual Care (Control) | Usual Care, Then PEGASUS Program (Intervention)
Number analyzed (Participants) | 263 | 242
mean percentage of guideline adherence
  Baseline, Isolated TBI (non-head AIS=0): number analyzed (Participants) | 20 | 19
  Baseline, Isolated TBI (non-head AIS=0) | 80.2 (12.1) | 84.3 (12.2)
  Baseline, Extracranial injury (non-head AIS>0): number analyzed (Participants) | 35 | 42
  Baseline, Extracranial injury (non-head AIS>0) | 83.0 (13.4) | 79.6 (13.4)
  Post-Randomization, Isolated TBI (non-head AIS=0): number analyzed (Participants) | 61 | 31
  Post-Randomization, Isolated TBI (non-head AIS=0) | 81 (13.9) | 86.2 (12.4)
  Post-Randomization, Extracranial injury (non-head AIS>0): number analyzed (Participants) | 147 | 150
  Post-Randomization, Extracranial injury (non-head AIS>0) | 84.8 (10.2) | 84.0 (12.9)
Statistical Analysis 1: Comparison: Usual Care, Then Usual Care (Control) vs Usual Care, Then PEGASUS Program (Intervention); Test type: Superiority; p = .01, Mixed Models Analysis — The outcome was analyzed using a multi-level mixed-effects model, which included a random effect for site (to account for potential provider clustering) and fixed effects for covariates; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 7.9, 95% CI 2-sided [1.9 to 13.8]

ADVERSE EVENTS:
Time Frame: Adverse events data (in-hospital complications and in-hospital mortality) were collected for all participants, all study periods (baseline and post-randomization), and all arms. Individual participants' data were collected for the timeframe of their study hospital admission date through their study hospital discharge which varied depending on the individual participant's clinical care needs and was not controlled by the study.
Description: Our in-hospital complications form reported pneumonia, arrhythmia, shock, peritonitis, intraparenchymal hemorrhages, and other complications as free text. Severity was reported as severe, moderate, or mild. Severe events are reported here as serious adverse events and moderate/mild as other adverse events. More than one complication, complication type, and severity could be reported for the same participant.
  Other was free text classified into organ system by investigators.
Groups:
- Usual Care at Baseline (Site That Was Later Assigned to the Control): All participants received Usual Care. This arm (8 sites) was randomized to maintain usual care (control) on 7/13/2020.
  Data for Adverse Events from the Baseline period (9/1/19-7/13/20) are listed here. See Outcomes for Mortality separated by study period.
- Usual Care at Post-Randomization Control Site: All participants received Usual Care. This arm (8 sites) was randomized to maintain usual care (control) on 7/13/2020.
  Data for Adverse Events from the Post-Randomization period (7/14/20-9/30/23) are listed here. See Outcomes for Mortality separated by study period.
  Sites will receive the opportunity for the PEGASUS program training (intervention) after the end of study.
- Usual Care at Baseline (Site That Was Later Assigned to the Intervention): All participants received Usual Care. This arm (8 sites) was randomized to PEGASUS (intervention) on 7/13/2020.
  Data for Adverse Events from the Baseline period (9/1/19-7/13/20) are listed here. See Outcomes for Mortality separated by study period.
- PEGASUS Program at Post-Randomization Intervention Site: All participants received the PEGASUS Program in addition to Usual Care. This arm (8 sites) was randomized to PEGASUS (intervention) on 7/13/2020.
  Data for Adverse Events from the Post-Randomization period (7/14/20-9/30/23) are listed here. See Outcomes for Mortality separated by study period.
  Intervention site training occurred before the intervention was implemented for participants admitted beginning 10/1/2020. Participants in the Post-Randomization were intention-to-treat once site arm was assigned. Participants in this study period received Usual Care while site were receiving pre-implementation training, after implementation, participants received Usual Care and the PEGASUS Program.
  See Outcomes for Mortality separated by study period.
  PEGASUS Program for Care: This is in essence a checklist of pediatric guidelines to follow for participants who meet inclusion criteria. Site staff will receive training in how to implement this pathway into their usual care.
Arm/Group | Usual Care at Baseline (Site That Was Later Assigned to the Control) | Usual Care at Post-Randomization Control Site | Usual Care at Baseline (Site That Was Later Assigned to the Intervention) | PEGASUS Program at Post-Randomization Intervention Site
All-Cause Mortality (participants affected / at risk) | 3/55 | 12/208 | 6/61 | 13/181
Serious Adverse Events (participants affected / at risk) | 6/55 | 34/208 | 7/61 | 17/181
Other Adverse Events (participants affected / at risk) | 21/55 | 72/208 | 16/61 | 78/181
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care at Baseline (Site That Was Later Assigned to the Control) (N=55) | Usual Care at Post-Randomization Control Site (N=208) | Usual Care at Baseline (Site That Was Later Assigned to the Intervention) (N=61) | PEGASUS Program at Post-Randomization Intervention Site (N=181)
Pneumonia (Infections and infestations) | 1 (1) | 9 (12) | 1 (1) | 5 (5) — Pneumonia, severe
Arrhythmia (Cardiac disorders) | 0 (0) | 2 (5) | 0 (0) | 1 (1) — Arrhythmia, severe
Shock (General disorders) | 4 (4) | 17 (23) | 3 (4) | 8 (8) — Shock, severe
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Peritonitis, severe
Intraparenchymal hemorrhage (Nervous system disorders) | 2 (2) | 3 (3) | 1 (1) | 2 (2) — Intraparenchymal hemorrhage, severe
Other: Respiratory (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 3 (3) | 2 (2) | 0 (0) — Other severe complications free text, classified by investigators as associated with Respiratory System
Other: Neurological (Nervous system disorders) | 0 (0) | 12 (15) | 1 (1) | 4 (10) — Other severe complications free text, classified by investigators as associated with Neurologic/Nervous System
Other: Electrolyte/Metabolic (Metabolism and nutrition disorders) | 0 (0) | 4 (9) | 0 (0) | 1 (2)
Other: Cardiac (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Other: Hematology (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Other: Infectious (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care at Baseline (Site That Was Later Assigned to the Control) (N=55) | Usual Care at Post-Randomization Control Site (N=208) | Usual Care at Baseline (Site That Was Later Assigned to the Intervention) (N=61) | PEGASUS Program at Post-Randomization Intervention Site (N=181)
Pneumonia (Infections and infestations) | 6 (7) | 49 (50) | 10 (11) | 40 (43) — Pneumonia, mild or moderate
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Arrhythmia, mild or moderate
Shock (General disorders) | 2 (3) | 3 (3) | 1 (1) | 2 (2) — Shock, mild or moderate
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) — Peritonitis, mild or moderate
Intraparenchymal hemorrhage (Nervous system disorders) | 2 (2) | 2 (2) | 1 (1) | 1 (1) — Intraparenchymal hemorrhage, mild or moderate
Other: Infectious (Infections and infestations) | 4 (5) | 4 (4) | 4 (4) | 19 (21) — Other mild or moderate complications free text, classified by investigators as associated with Infections
Other: Respiratory (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 4 (4) | 0 (0) | 3 (3) — Other mild or moderate complications free text, classified by investigators as associated with Respiratory System
Other: Neurological (Nervous system disorders) | 5 (7) | 20 (22) | 2 (3) | 21 (24) — Other mild or moderate complications free text, classified by investigators as associated with Neurologic/Nervous System
Other: Gastrointestinal (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) — Other mild or moderate complications free text, classified by investigators as associated with Gastrointestinal System
Other: Hematology (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 1 (1) | 3 (3) — Other mild or moderate complications free text, classified by investigators as associated with Hematology
Other: Cardiac (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Other mild or moderate complications free text, classified by investigators as associated with Cardiology
Other: Electrolyte/Metabolic (Metabolism and nutrition disorders) | 1 (1) | 2 (3) | 1 (1) | 2 (2) — Other mild or moderate complications free text, classified by investigators as associated with Electrolytes/Metabolic
Other: Ophthalmalogical (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) — Other mild or moderate complications free text, classified by investigators as associated with Ophthalmology
Other: Kidney (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Other mild or moderate complications free text, classified by investigators as associated with Kidney/Nephrology
Other: Dermatological (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Other mild or moderate complications free text, classified by investigators as associated with Dermatology

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-08-07): https://cdn.clinicaltrials.gov/large-docs/89/NCT03896789/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-10): https://cdn.clinicaltrials.gov/large-docs/89/NCT03896789/SAP_001.pdf
  • Informed Consent Form (2019-08-15): https://cdn.clinicaltrials.gov/large-docs/89/NCT03896789/ICF_002.pdf